CLINICAL TRIAL: NCT05478096
Title: The Caring Universities Project: RCT Evaluating the Effectiveness of a Guided E-health Programme (GetStarted) in Reducing Procrastination in University Students
Brief Title: The Caring Universities Project: GetStarted RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: VU University of Amsterdam (Other)
Collaborators: Leiden University (Other); Maastricht University (Other); Utrecht University (Other); Erasmus University Rotterdam (Other)
Responsible Party: Principal Investigator, Arpana Amarnath, Associate researcher, VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VCWE-2021-193
Record Dates: First submitted 2022-07-25; First posted 2022-07-28 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Procrastination
Keywords: procrastination; guided; e-health; university students; mental health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The present study is a two-arm randomized control superiority trial. This trial will be conducted in a university setting. A guided web-based anti-procrastination programme (GetStarted) will be compared to a waiting list condition.
Who Masked: Investigator, Outcomes Assessor
Masking Description: An independent researcher who is not involved in the study will generate the random sequence using a computer random sequence generator. Randomisation will take place at an individual level, stratified by gender and the university where students study. Participants will be randomised into two groups (web-based intervention vs. WL) with allocation ratio of 1:1. We will conduct block randomisation with randomly varied block sizes (6 to 12 allocations per block) to prevent foreknowledge of intervention assignment. Allocation will be concealed from the study's researchers. It is not possible to mask personnel and participants to the treatment allocation because of the nature of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- We-based intervention for procrastination (Experimental): GetStarted is a guided e-health application, based on cognitive-behavioral therapy (CBT). It comprises 5 main and 4 optional modules that are delivered weekly via computer, laptop, tablet, or mobile phone. Every week a trained e-coach will provide feedback on the progress of the program and the exercises via e-mail. The main modules are (1) psycho-education about procrastination (2) getting insight into one's own procrastination behavior, (3) uncovering unhelpful thoughts underlying procrastination and (4) replacing these unhelpful thoughts with helpful ones. Each module takes approximately 40 minutes to complete and participants will receive provide asynchronous written personalized feedback from their e-coaches within 48 hours (counting workdays only) after session completion.
  Interventions: Behavioral: GetStarted
- Wait list (No Intervention): Participants in the waiting list condition will receive no treatment for four weeks post-randomization. Following this, they can start the program if they choose to do so.

INTERVENTIONS:
Behavioral: GetStarted — Guided internet-based intervention for procrastination.
  Arms: We-based intervention for procrastination

SUMMARY:
Within the Caring Universities project (study protocol VCWE- 2020-076 accepted by the VCWE), we have developed a guided e-health programme (GetStarted) designed to reduce procrastination in university students. With the current study, we aim to examine the effectiveness of GetStarted in reducing procrastination behaviour. Secondary goals are to gain an insight into pre-test to post-test differences regarding symptoms of low mood, anxiety and quality of life. Additionally, we aim to gain insight into the effects of participants' satisfaction with the intervention and Ecoach, the usability of the program, and treatment adherence on the effectiveness of the treatment.

DETAILED DESCRIPTION:
The present study is a two-arm randomized control superiority trial. This trial will be conducted in a university setting. A guided web-based anti-procrastination programme (GetStarted) will be compared to a waiting list condition.

GetStarted was developed based on existing literature and adapted in collaboration with university students to meet the specific needs of the university students. We have conducted interviews with students to understand their opinions about this program and adapted it based on their preferences and needs. The programme is based on cognitive-behavioral therapy (CBT). It comprises five main modules that are delivered via computer, laptop, tablet, or mobile phone and four optional modules. Every module consists of evidence-based information, exercises, and homework assignments. The content is delivered in text format with pictures and infographics; some modules also include video clips and audio recordings on a relevant subject. The intervention is available in both English and Dutch.

Every week trained e-coaches (trained clinical psychology master students) will provide asynchronous written personalized feedback to each participant on the progress of the program and the exercises via the program platform. Measurements include pre- and post-assessment of procrastination behavior, common measures of psychopathology symptoms, quality of life, treatment adherence, program usability and participants' satisfaction with treatment and coaching.

All students currently enrolled at the participating universities (Vrije Universiteit Amsterdam, Erasmus University, Universities of Leiden, Utrecht and Maastricht) are potentially eligible for the trial.

Benefits of participation and remuneration for the test subjects:

Students can participate in GetStarted free of charge, which will likely decrease their procrastination behavior. They do not receive any monetary incentives.

ELIGIBILITY:
Inclusion Criteria:

* aged 16 or older
* enrolled at one of the participating universities
* fluent in Dutch and/or English
* access to a PC or mobile device with internet access
* score 32 or above on the Irrational Procrastination Scale (IPS)
* provide informed consent.

Exclusion Criteria:

* any suicidal risk by identifying if they (the participants) have had thoughts of killing themselves or have made plans of killing themselves in the past year and then responding to the question "How likely do you think it is that you will act on this plan in the next 12 months?" with somewhat likely or very likely

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2021-11-19 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Change in procrastination behaviours | T0/T1 (Baseline) to T2/T3 (Post-test: 4-weeks) to T5 (Follow up: 6 months)
  The Irrational Procrastination Scale (IPS) is used to assess procrastination tendencies by assessing extent to which participants procrastinate. This scale contains 9 items scored on a five-point Likert scale ranging from 1 (very seldom or not true to me) to 5 (very often true or true to me).The total scores can range from 9 to 45 with highers score indicating higher levels of procrastination.

SECONDARY OUTCOMES:
Change in depressive symptoms | T1 (Baseline) to T2/T3 (Post-test: 4-weeks) to T5 (Follow up: 6 months)
  The Patient Health Questionnaire (PHQ-9) is used as the measure of depression. This questionnaire consists of 9 items scored on a four-point Likert scale ranging from 0 (not at all) to 3 (nearly every day). The total scores can range from 0 to 27, with higher scores indication more severe depressive symptoms
Change in severity of stress | T1 (Baseline) to T2/T3 (Post-test: 4-weeks) to T5 (Follow up: 6 months)
  The perceived stress scale (PSS-10) is used as a self-report measure of perceived stress. It consists of 10 items scored on a five-point Likert scale ranging from 0 (never) to 4 (very often). The total scores range from 0-40, with a higher score indicating higher levels of perceived stress.
Change in quality of life | T1 (Baseline) to T2/T3 (Post-test: 4-weeks) to T5 (Follow up: 6 months)
  The Mental Health Quality of Life questionnaire (MHQoL) is used to measure quality of life. It consists of 7 items scored on a four-point Likert scale ranging from 0 (very dissatisfied) to 3 (very satisfied). The total scores can range from 0-21 with higher scores indicating better quality of life.
Change in Anxiety symptoms | T1 (Baseline) to T2/T3 (Post-test: 4-weeks) to T5 (Follow up: 6 months)
  The Generalized Anxiety Disorder scale (GAD-7) is used to measure symptoms of generalized anxiety. The questionnaire consists of 7 items measured on a four-point Likert ranging from 0 (not at all) to 3 (nearly every day). The total scores range from 0 to 21 with higher scores indicating more severe GAD symptoms.

OTHER OUTCOMES:
Socio demographic characteristics and additional participant information | T0 (Baseline)
  * age
  * gender
  * ethnicity
  * student status
  * study level
  * relationship status
  * whether the student is currently undergoing any treatment (pharmacotherapy/psychotherapy/both/none)
Satisfaction with the intervention | T2 (Post-test: 4-weeks)
  The Client Satisfaction Questionnaire (CSQ-8) is used to measure participants' satisfaction with the overall intervention. The CSQ-8 is commonly used to measure satisfaction with online interventions. It consists of eight items on a four-point Likert scale with a total score ranging from 8 to 32, where a higher score indicates greater satisfaction.
Usability | T2 (Post-test: 4-weeks)
  The System Usability Scale (SUS-10) is used to measure the usability of the intervention. It consists of 10 items on a five-point Likert scale with a total score ranging from 0 to 100, where a higher score indicates greater usability.
Adherence | T2 (Post-test: 4-weeks)
  Adherence refers to "the degree to which the user followed the program as it was designed" (Donkin et al., 2011). The present study measures adherence by dividing the number of modules completed by a participant at time of post-test by the total number of modules in the programme, and multiplying this by 100. The resulting percentage will indicate completion rate.
Satisfaction with E-coach | T2 (Post-test: 4-weeks)
  The Working Alliance Inventory for guided internet interventions (WAI-I) is used to evaluate participant's satisfaction with the e-coach. The WAI-I consists of 12 items on a 5-point Likert scale with a total score ranging from 12 to 60, where higher scores indicate higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Y Struijs, PhD, Principal Investigator — VU University of Amsterdam
Locations (1):
- Vrije Universiteit Amsterdam, Amsterdam, Netherlands

REFERENCES:
- [Derived] Amarnath A, Ozmen S, van Klaveren C, van Straten A, Pei J, de Wit L, Raabe RE; Caring Universities Consortium; Cuijpers P, Struijs SY. Effectiveness of a guided internet-based intervention in reducing procrastination among university students - a randomized controlled trial. Internet Interv. 2025 Sep 29;42:100878. doi: 10.1016/j.invent.2025.100878. eCollection 2025 Dec. PMID 41080972
- [Derived] Amarnath A, Ozmen S, Struijs SY, de Wit L, Cuijpers P. Effectiveness of a guided internet-based intervention for procrastination among university students - A randomized controlled trial study protocol. Internet Interv. 2023 Mar 3;32:100612. doi: 10.1016/j.invent.2023.100612. eCollection 2023 Apr. PMID 36922962